CLINICAL TRIAL: NCT00219167
Title: An 8-week, Randomized, Double-blind, Parallel-group, Multicenter Study Assessing the Efficacy and Safety of Aliskiren 75 mg, 150 mg, and 300 mg in Patients With at Least 65 Years of Age With Essential Hypertension, Using 24-hour ABPM, With Lisinopril 10 mg as a Reference
Brief Title: A Clinical Study to Assess Efficacy and Safety of Aliskiren in the Elderly With High Blood Pressure
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CSPP100A2324
Record Dates: First submitted 2005-09-12; First posted 2005-09-22 (Estimated); Last update posted 2016-11-18 (Estimated); Status verified 2016-11

CONDITIONS: Hypertension
Keywords: hypertension; aliskiren; age
MeSH Terms: conditions — Hypertension | interventions — aliskiren

INTERVENTIONS:
Drug: aliskiren

SUMMARY:
After a wash-out (1 to 2 weeks), and 2 to 4 week single-blind placebo run-in period, eligible patients will be randomized to receive lisinopril 10 mg, aliskiren 75 mg, 150 mg or 300 mg for a period of 8 weeks

ELIGIBILITY:
Inclusion Criteria

* Patients with at least 65 years-old
* Patients with essential hypertension Exclusion Criteria
* Severe hypertension
* History or evidence of a secondary form of hypertension
* History of Hypertensive encephalopathy or cerebrovascular accident. Other protocol-defined inclusion exclusion criteria also apply.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 355 (Actual)
Dates: Start 2005-04; Primary Completion 2006-02 (Actual); Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
Change from baseline in average 24 hour systolic ambulatory blood pressure after 8 weeks

SECONDARY OUTCOMES:
Change from baseline in average 24 hour diastolic ambulatory blood pressure after 8 weeks
Change from baseline in sitting systolic and diastolic blood pressure after 8 weeks
Change from baseline in daytime diastolic ambulatory blood pressure after 8 weeks
Change from baseline in daytime systolic ambulatory blood pressure after 8 weeks
Blood pressure control target of < 140/90 mmHg after 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Pharmaceuticals, Basel, Switzerland

REFERENCES:
- [Result] Verdecchia P, Calvo C, Mockel V, Keeling L, Satlin A. Safety and efficacy of the oral direct renin inhibitor aliskiren in elderly patients with hypertension. Blood Press. 2007;16(6):381-91. doi: 10.1080/08037050701717014. PMID 18058456
- [Derived] Wang GM, Li LJ, Tang WL, Wright JM. Renin inhibitors versus angiotensin converting enzyme (ACE) inhibitors for primary hypertension. Cochrane Database Syst Rev. 2020 Oct 22;10(10):CD012569. doi: 10.1002/14651858.CD012569.pub2. PMID 33089502